CLINICAL TRIAL: NCT03138538
Title: An Open-label, Phase I Dose Escalation Trial of Methionine Aminopeptidase 2 Inhibitor M8891 in Subjects With Advanced Solid Tumors
Brief Title: M8891 First in Human in Solid Tumors
Acronym: M8891
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: As part of a portfolio-level management of the company's oncology pipeline, it was decided to stop the next phase of internal development of the MetAP2 (M8891) program to enable realization of other opportunities within the oncology portfolio.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS100015_0019
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumors; Metastatic Renal Cell Carcinoma
Keywords: Advanced Solid Tumors; Metastatic Renal Cell Carcinoma; M8891; Methionine Aminopeptidase 2 Inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- M8891 7 mg (Experimental): Participant received M8891 at dose of 7 milligrams (mg) orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Interventions: Drug: Part 1: M8891
- M8891 12 mg (Experimental): Participant received M8891 at dose of 12 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Interventions: Drug: Part 1: M8891
- M8891 20 mg (Experimental): Participant received M8891 at dose of 20 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Interventions: Drug: Part 1: M8891
- M8891 35 mg (Experimental): Participant received M8891 at dose of 35 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Interventions: Drug: Part 1: M8891
- M8891 60 mg (Experimental): Participant received M8891 at dose of 60 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Interventions: Drug: Part 1: M8891
- M8891 80 mg (Experimental): Participant received M8891 at dose of 80 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Interventions: Drug: Part 1: M8891

INTERVENTIONS:
Drug: Part 1: M8891 — Participants receives M8891 orally once daily at escalated dose levels under fasting condition for consecutive 21-day cycles of continuous treatment until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose (MTD), safety, tolerability, Pharmacokinetic (PK), pharmacodynamic and clinical activity of M8891 as single agent in participants with advanced solid tumors in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be refractory to or intolerant of existing cancer therapy(ies) known to provide clinical benefit.
* Histologically confirmed advanced solid tumors with no clear curative treatment options available after at least 1 prior systemic anticancer therapy.
* Tumor accessible for biopsies and agreement to conduct pre-dose and post-dose fresh tumor biopsies.
* Male or female subjects at least 18 years of age
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at Screening
* Histologic or cytologic evidence/proven of metastatic renal cell carcinoma (mRCC) with clear cell component
* Part 2A: Participants should have progressed to 1 or more previous lines of systemic anticancer therapy, excluding treatment with cabozantinib
* Part 2B: Participants should have progressed to 1 or 2 previous lines of systemic anticancer therapy, excluding treatment with cabozantinib. Participants should have failed to only 1 previous TKI for metastatic disease. Adjuvant therapy with sunitinib will be considered as 1 line of therapy for metastatic disease in the case that disease progression occurs during or within 3 months of the completion of the treatment.
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* ECOG PS >= 2
* Extensive prior radiotherapy on more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation within 5 years of study start.
* Severe bone marrow, renal or liver impairment.
* Tumor in contact with, invading or encasing major blood vessels or radiographic evidence of significant cavitary pulmonary lesions
* Uncontrolled hypertension defined as sustained Blood Pressure (BP) > 150 millimeters of mercury (mm Hg) systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment
* Participant is pregnant or breastfeeding
* Part 2A and 2B: Previous use of cabozantinib or a MetAP2 inhibitor, tumor in contact with invading or encasing major blood vessels or radiographic evidence of significant cavitary pulmonary lesions
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (7):
- United States (7):
  - Smilow Cancer Hospital - Yale, New Haven, Connecticut
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Sidney Kimmel Cancer Center - Johns Hopkins, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- [Derived] Lignet F, Friese-Hamim M, Jaehrling F, El Bawab S, Rohdich F. Preclinical Pharmacokinetics and Translational Pharmacokinetic/Pharmacodynamic Modeling of M8891, a Potent and Reversible Inhibitor of Methionine Aminopeptidase 2. Pharm Res. 2023 Dec;40(12):3011-3023. doi: 10.1007/s11095-023-03611-z. Epub 2023 Oct 5. PMID 37798538
- [Derived] Carducci MA, Wang D, Habermehl C, Bodding M, Rohdich F, Lignet F, Duecker K, Karpenko O, Pudelko L, Gimmi C, LoRusso P. A First-in-human, Dose-escalation Study of the Methionine Aminopeptidase 2 Inhibitor M8891 in Patients with Advanced Solid Tumors. Cancer Res Commun. 2023 Aug 24;3(8):1638-1647. doi: 10.1158/2767-9764.CRC-23-0048. eCollection 2023 Aug. PMID 37637935
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100015_0019
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): 08 August 2017. Last participant completed: 16 September 2020.
Pre-assignment Details: This study was to be conducted in 2 parts; Part 1 was the dose escalation phase and Part 2 was the expansion phase. However, due to early termination of the study, the sponsor decided not to conduct the expansion phase (Part 2).
Period: Overall Study
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Started | 3 | 3 | 3 | 8 | 7 | 3
Completed | 3 | 3 | 3 | 8 | 7 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- M8891 7 mg: Participant received M8891 at dose of 7 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
- Total: Total of all reporting groups
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 4 | 3 | 0 | 14
  >=65 years | 1 | 0 | 1 | 4 | 4 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 3 | 3 | 2 | 13
  Male | 0 | 2 | 2 | 5 | 4 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 0 | 2
  White | 2 | 3 | 3 | 4 | 6 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs) Assessed Using National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03
Description: A DLT was defined as the occurrence of any of following events that were judged by the study investigator, to be related to the study medication: Grade 4 liver enzyme elevation; Grade 4 neutropenia lasting >5 days or Grade >= 3 neutropenia with fever; Grade 4 thrombocytopenia lasting >5 days or Grade >=3 thrombocytopenia with clinically significant bleeding; Any treatment interruption >7 days or >30% of total dose in Cycle 1 due to AEs not related to the underlying disease or concomitant medication; Grade >=3 non-hematologic toxicity excluding Grade 3 nausea or vomiting lasting <48 hours, and resolves to <= Grade 1 either spontaneously or with medication, Grade 3 fatigue <= 3 days, Grade 3 hypertension in the absence of maximal medical therapy, Grade 3 rash <= 3 days, Grade 3 electrolyte abnormality that lasts <72 hours, is not clinically complicated, and resolves spontaneously or responds to conventional medication and Grade >=3 single lab value increase without clinical correlate.
Time Frame: At the end of Cycle 1 (each Cycle is of 21 days)
Population: Dose escalation set included all participants treated in dose-escalation cohorts who did not miss > 4 cumulative days planned doses of M8891 in the first cycle of the dose-escalation part for other than safety reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 2 | 5 | 5 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 1

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) and TEAEs Leading to Death
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- M8891 80 mg: Participant received M8891 at dose of 12 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants
  TEAEs | 3 | 2 | 3 | 8 | 7 | 3
  TEAEs leading to death | 0 | 1 | 2 | 2 | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) by Severity
Description: Severity of adverse events (AE) were assessed by the investigator according to National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03 as Grade 1 to Grade 5. Grade 1= Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4= Life-threatening and Grade 5= Death. The number of participants that experienced at least one solicited local TEAE were summarized by grade. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs. Number of participants with Grade >=3, >=4 and 5 were reported.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants
  Grade >=3 | 0 | 1 | 3 | 8 | 4 | 2
  Grade >=4 | 0 | 1 | 2 | 2 | 1 | 1
  Grade 5 | 0 | 1 | 2 | 2 | 0 | 0

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of M8891
Description: Maximum observed plasma concentration (Cmax) was taken directly from the observed concentration-time curve.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: Pharmacokinetic (PK) analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. Here "Number Analyzed"=number of participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Nanogram per milliliter (ng/mL)
  Day 1 | 514 (16.6) | 934 (12.4) | 1780 (48.9) | 2960 (17.0) | 3630 (31.2) | 4760 (15.6)
  Day 15: number analyzed (Participants) | 3 | 3 | 2 | 5 | 4 | 2
  Day 15 | 1260 (39.2) | 2210 (21.1) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values. | 6840 (16.9) | 6600 (20.2) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values.

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of M8891
Description: The time to reach the maximum observed plasma concentration (tmax) was obtained directly from the concentration versus time curve.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: PK analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. Here "Number Analyzed"=number of participants evaluable at specified time points.
Measure: Median (Full Range); unit: Hour
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Hour
  Day 1 | 3.17 [3.00 to 24.0] | 4.00 [2.00 to 11.0] | 6.00 [2.23 to 6.73] | 4.04 [2.92 to 8.02] | 7.13 [4.12 to 23.9] | 3.38 [1.87 to 8.07]
  Day 15: number analyzed (Participants) | 3 | 3 | 2 | 5 | 4 | 3
  Day 15 | 4.00 [3.10 to 4.98] | 2.00 [1.10 to 3.00] | NA [2.83 to 3.97] — Based on pre-specified criteria Median was not calculated if fewer than 3 participants have reportable parameter values. | 4.07 [1.32 to 8.00] | 3.11 [2.05 to 22.8] | NA [1.98 to 4.18] — Based on pre-specified criteria Median was not calculated if fewer than 3 participants have reportable parameter values.

6. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of M8891
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification (LLOQ), calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Nanogram*hour per milliliter (ng*h/mL)
  Day 1 | 9080 (21.3) | 16300 (9.6) | 34200 (41.0) | 59400 (22.7) | 71700 (26.3) | 86900 (22.5)
  Day 15: number analyzed (Participants) | 3 | 3 | 2 | 5 | 4 | 2
  Day 15 | 25400 (50.3) | 38600 (17.6) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values. | 141000 (13.9) | 134000 (18.4) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values.

7. Secondary Outcome: Area Under the Concentration-time Curve From Zero Extrapolated to Infinity (AUC0-inf) of M8891
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from the determination of the terminal first order (elimination) rate constant (lambda z). AUC0-inf = AUC0-t plus Clast pred/lambda z. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve. Clastpred was the last predicted quantifiable concentration.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: PK analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. As R2 was <0.80, %AUCextra was >20% and elimination phase was not characterized, AUC0-inf derived from lambda z was regarded as implausible and not calculated.
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Within One Dosing Interval (AUC0-tau) of M8891
Description: AUC (0-tau) is the area under the plasma concentration time curve within 1 dosing interval. Calculated using the mixed log linear trapezoidal rule (linear up, log down).
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
ng*h/mL
  Day 1 | 9100 (21.2) | 16300 (9.6) | 32400 (35.7) | 59100 (20.3) | 71400 (26.8) | 84500 (20.6)
  Day 15: number analyzed (Participants) | 3 | 3 | 2 | 5 | 4 | 2
  Day 15 | 25700 (48.4) | 38500 (18.7) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values. | 137000 (15.6) | 133000 (17.4) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values.

9. Secondary Outcome: Apparent Terminal Half Life (t1/2) of M8891
Description: Terminal half-life of M8891 in Plasma was calculated as log2/ lambda z. Lambda z was determined from the terminal slope of the log-transformed concentration curve using linear regression on terminal data points of the curve.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: PK analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. As coefficient of correlation (R2) was <0.80, %AUCextra was >20% and elimination phase was not characterized, t1/2 derived from lambda z was regarded as implausible and not calculated.
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Terminal Elimination Rate Constant (Lambda z) of M8891
Description: Lambda z was determined from the terminal slope of the log-transformed concentration curve using linear regression on terminal data points of the curve.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: PK analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. As R2 was <0.80, %AUCextra was >20% and elimination phase was not characterized, lambda z was regarded as implausible and not calculated.
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Apparent Total Body Clearance (CL/f) of M8891
Description: Apparent total body clearance of drug from plasma following extravascular administration, calculated as dose/AUC0-infinity for M8891. Area under the plasma concentration-time curve from time zero (dosing time) extrapolated to infinity of unchanged drug calculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-infinity calculated by Clastpred/lambda z, where Clastpred is the predicted plasma concentration at the last sampling time point, calculated from the log linear regression line for lambda z determination at which the measured plasma concentration is at or above lower limit of quantification.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: PK analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. As R2 was <0.80, %AUCextra was >20% and elimination phase was not characterized, CL/f derived from lambda z was regarded as implausible and not calculated.
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Apparent Body Clearance of Drug Following Extravascular Administration At Steady State (CLss/f) of M8891
Description: The apparent total body clearance of drug at steady state following extravascular administration, taking into account the fraction of dose absorbed. It is calculated as dose/AUCtau for M8891.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: PK analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. As R2 was <0.80, %AUCextra was >20% and elimination phase was not characterized, CLss/f derived from lambda z was regarded as implausible and not calculated.
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (VZ/f) of M8891
Description: Apparent volume of distribution during the terminal phase following extravascular administration for M8891 was calculated. Vz/f = Dose/(AUC0-infinity multiply by Lambda z) following single dose. The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination. AUC(0- inf)=AUC0-t plus Clastpred/lambda z where Clastpred was last predicted concentration. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: Cycle 1 Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 (Each cycle is of 21 days)
Population: PK analysis set included all participants from the safety analysis set without major protocol deviations/violations or events that would affect PK. As R2 was <0.80, %AUCextra was >20% and elimination phase was not characterized, VZ/f derived from lambda z was regarded as implausible and not calculated.
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Accumulation Ratios of AUC (Racc AUC) of M8891
Description: Racc (AUC) is defined as the accumulation factor to assess the increase in exposure until steady state is reached. Accumulation ratio for AUC was calculated as AUC, after dosing on Day 15 divided by AUC, after dosing on Day 1 of Cycle 1.
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 of Cycle 1 (each cycle is 21 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 2 | 5 | 4 | 2
Ratio | 2.82 (29.3) | 2.36 (27.4) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values. | 2.38 (27.8) | 1.90 (37.2) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values.

15. Secondary Outcome: Accumulation Ratio of Cmax (Racc Cmax) of M8891
Description: Accumulation ratio of Cmax was calculated as Cmax, after dosing on Day 15 divided by Cmax, after dosing on Day 1 of Cycle 1.
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose on Day 1 and 15 of Cycle 1 (each cycle is 21 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 2 | 5 | 4 | 2
Ratio | 2.46 (27.5) | 2.36 (33.5) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values. | 2.32 (27.4) | 1.97 (37.8) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values.

16. Secondary Outcome: Number of Participants With Best Overall Response Assessment According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: BOR was determined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as assessed by investigators. BOR is defined as the best response of any of the complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from the date of randomization until disease progression. CR: Disappearance of all evidence of target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD) defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD while on study. PD is defined as at least a 20 percent (%) increase in the SLD of target lesion, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 2 | 2 | 1 | 0 | 2 | 0
  Progressive Disease | 1 | 0 | 0 | 3 | 1 | 1
  Not Evaluable | 0 | 1 | 2 | 5 | 4 | 2

17. Secondary Outcome: Number of Participants With Clinical Benefit
Description: Clinical benefit defined as Complete Response (CR), Partial Response (PR) or Stable Disease (SD) for >= 12 weeks. Clinical benefit was assessed according to RECIST Version 1.1. CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest SLD while on study. PD is defined as at least a 20 percent (%) increase in the SLD of target lesion, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 2 | 0 | 0 | 0 | 1 | 0

18. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) defined as the time from first study drug administration to either first observation of progressive disease (PD) (as assessed by Investigators according to RECIST v1.1) or occurrence of death due to any cause, whichever occurs first. Progressive disease (PD) defined as at least a 20% increase in sum of longest diameter (SLD) of target lesions, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier (KM) estimates. Here the 20 mg dose level was selected for stratification as the highest dose level equal to or smaller than the median of all dose levels administered to at least 1 participant.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Less Than or Equal to (<=) 20 mg M8891: All participants who received oral capsule of M8891 at dose <= 20 mg first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
- Greater Than (>) 20 mg M8891: All participants who received oral capsule of M8891 at dose of > 20mg first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
Arm/Group | Less Than or Equal to (<=) 20 mg M8891 | Greater Than (>) 20 mg M8891
Number analyzed (Participants) | 9 | 18
Months | 2.7598 [1.05 to 4.40] | 1.3799 [0.82 to 1.54]

19. Secondary Outcome: Number of Participants With Change From Baseline in Laboratory Test Abnormalities to Grade 3 or Higher Severity Based on NCI-CTCAE Version 4.03
Description: The laboratory measurements included hematology, biochemistry, and urinalysis values were graded with National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 toxicity grades (where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = death). Number of participants with change from baseline to grade 3 or higher values for the hematology, biochemistry and urinalysis parameters were reported.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- M8891 12 mg qd: Participant received M8891 at dose of 12 mg orally with first dose in Cycle 1 Day 1 and consist of consecutive 21-day cycles of continuous once daily M8891 monotherapy under fasting conditions until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
Arm/Group | M8891 7 mg | M8891 12 mg qd | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants
  Grade >= 3 biochemistry | 0 | 0 | 2 | 2 | 3 | 0
  Grade >= 3 hematology | 0 | 0 | 1 | 2 | 4 | 1
  Grade >= 3 urinalysis | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Vital Signs
Description: Vital sign assessments included assessments of heart rate, diastolic blood pressure, systolic blood pressure, weight, respiratory rate and temperature. Clinical relevance was assessed by the investigator. Number of participants who had any clinically meaningful change from baseline in vital signs were reported.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Electrocardiogram (ECG) Values
Description: ECG parameters included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, QT intervals, and corrected QT(QTc) intervals. Clinical significance was determined by the investigator. Number of participants with clinically meaningful change from baseline in 12-lead ECG were reported.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PF) Score of 2 or Higher Than 2
Description: ECOG PS score is widely used by doctors and researchers to assess how a participants' disease is progressing, and is used to assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. The score ranges from Grade 0 to Grade 5, where Grade 0 = Fully active, able to carry on all pre-disease performance without restriction, Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (like light house work, office work), Grade 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, Grade 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours and Grade 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair, Grade 5 = Death. Number of participants with ECOG performance status score of 2 or higher than 2 were reported.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Participants | 0 | 1 | 1 | 1 | 0 | 0

23. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response is defined as the percentage of participants with complete response (CR) and partial response (PR). CR is defined as disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions.
Time Frame: Up to 1136 Days
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
Number analyzed (Participants) | 3 | 3 | 3 | 8 | 7 | 3
Percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 60.2] | 0 [0.0 to 52.2] | 0 [0.0 to 97.5]

ADVERSE EVENTS:
Time Frame: Up to 1136 Days
Arm/Group | M8891 7 mg | M8891 12 mg | M8891 20 mg | M8891 35 mg | M8891 60 mg | M8891 80 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 2/3 | 2/8 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 3/3 | 3/8 | 1/7 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 8/8 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M8891 7 mg (N=3) | M8891 12 mg (N=3) | M8891 20 mg (N=3) | M8891 35 mg (N=8) | M8891 60 mg (N=7) | M8891 80 mg (N=3)
Disease progression (General disorders) | 0 | 1 | 2 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M8891 7 mg (N=3) | M8891 12 mg (N=3) | M8891 20 mg (N=3) | M8891 35 mg (N=8) | M8891 60 mg (N=7) | M8891 80 mg (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 3 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 3 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 4 | 2 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 2 | 5 | 2
Weight decreased (Investigations) | 0 | 0 | 2 | 2 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 2 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 3 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03138538/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03138538/SAP_001.pdf